CLINICAL TRIAL: NCT05343091
Title: Prognostic Value of the Evaluation of Right Ventricular Function by Portable Ultrasound in Patients With Pulmonary Hypertension.
Brief Title: Prognostic Value of the Right Ventricular Function by Portable Ultrasound in Patients With Pulmonary Hypertension.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: Pamela Mercado Velázquez (Unknown); Consuelo Orihuela Sandoval (Unknown); Tatiana Sofia Rodríguez Reyna (Unknown); Ivette Buendía Roldán (Unknown)
Responsible Party: Principal Investigator, Jose Luis Hernandez Oropeza, PhD, Head of Cardiopneumology Department, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Other Study IDs: 3492
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Pulmonary Hypertension; Pulmonary Arterial Hypertension; Cardiac Ultrasound
Keywords: Pulmonary hypertension; cardiac ultrasound; tricuspid annular plane systolic excursion; pulmonary arterial hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pulmonary Hypertension patients: patients with diagnosis of Pulmonary Hypertension from group 1 and 4 by right heart catheterization
  Interventions: Device: cardiac ultrasound

INTERVENTIONS:
Device: cardiac ultrasound — Cardiac ultrasound with Pocket ultrasound by expert and non expert physician

SUMMARY:
Pulmonary arterial hypertension (PAH) is a disease characterized by obliteration and remodeling of small-caliber pulmonary arteries, progressively generating an increase in pulmonary vascular resistance, right heart failure, and death. Current guidelines recommend a multidimensional approach which includes clinical, echocardiographic, exercise and hemodynamic variables to classify patients by risk and thus define a prognosis and guide therapeutic decisions.

There is a wide range of studies, which have shown a good correlation between standard echocardiography and portable cardiac ultrasound. There is no doubt about the usefulness of portable cardiac ultrasound in the intensive care unit, emergency department and even during hospital rounds; however, its usefulness during the daily examination in a follow-up consultation of patients at high risk of cardiovascular deterioration, such as patients with PAH, has not yet been demonstrated.

There is evidence that a TAPSE measurement <17mm using standard echocardiography by a physician experienced in echocardiography predicts survival in patients with Pulmonary hypertension. We would like to know if patients with low TAPSE will have a higher proportion of morbidity events compared to patients with normal TAPSE measured by portable ultrasound.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a disease characterized by obliteration and remodeling of small-caliber pulmonary arteries, progressively generating an increase in pulmonary vascular resistance, right heart failure, and death. Current guidelines recommend a multidimensional approach which includes clinical, echocardiographic, exercise and hemodynamic variables to classify patients by risk and thus define a prognosis and guide therapeutic decisions.

Transthoracic Echocardiography (TTE) currently plays an important role in the diagnostic algorithm of PAH as it is minimally invasive and readily available. Moreover, many echocardiographic parameters are closely related to pulmonary hemodynamics. Some TTE parameters are associated with mortality and surviving in these patients, such as: shortening fraction, presence of pericardial effusion, eccentricity index, systolic displacement of the tricuspid annular plane (TAPSE), size of the right atrium and right ventricular free wall strain.

Ultrasound (US) is the only method which enables realtime bedside imaging of the heart. Focused cardiac US provides worthy diagnostic information useful for the the clinical management of critical care patients. The use of cardiac ultrasound in the last decade has gradually increased among non cardiologists. Pocket ultrasounds are part of the third generation of ultrasounds described in the literature. These have the characteristic of being light devices weighing less than 1kg and that can be carried in the pocket of the medical uniform. This leads many researchers to believe that in the not too distant future its use will be part of the physical examination routine, as the stethoscope is now.

There is a wide range of studies, which have shown a good correlation between standard echocardiography and portable cardiac ultrasound. There is no doubt about the usefulness of portable cardiac ultrasound in the intensive care unit, emergency department and even during hospital rounds; however, its usefulness during the daily examination in a follow-up consultation of patients at high risk of cardiovascular deterioration, such as patients with PAH, has not yet been demonstrated.

STATEMENT OF THE PROBLEM Does the measurement of tricuspid annular plane systolic displacement (TAPSE) by portable cardiac ultrasound have prognostic utility in the follow-up of patients with Pulmonary Hypertension?

JUSTIFICATION There is evidence that a TAPSE measurement <17mm using standard echocardiography by a physician experienced in echocardiography predicts survival in patients with Pulmonary hypertension. However, the high costs of an apparatus to perform the standard echocardiogram study and the prolonged appointments to perform the study delay the diagnosis of treatment of progression of cardiovascular disease. Therefore, it is important to document the usefulness of using an accessible medical tool during the cardiopulmonology consultation for the follow-up of patients with pulmonary hypertension.

HYPOTHESIS Patients with low TAPSE will have a higher proportion of morbidity events compared to patients with normal TAPSE.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of Pulmonary Hypertension group 1 and 4 by right heart catheterization.
* Presence of a baseline transthoracic echocardiogram as well as a follow-up echocardiogram.
* Presence of 6m baseline walk as well as follow-up.

Exclusion Criteria:

* All patients with left heart disease associated with PH
* All patients with pulmonary disease associated with PH
* All patients with congenital heart disease who had poor surgical repair.
* Patients who meet the contraindication by the American chest guidelines to perform the 6m walk test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the diagnosis of Pulmonary Hypertension group 1 and 4 by right heart catheterization.
Sampling Method: Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
morbidity events with TAPSE | 9 months
  Estimate the risk of morbidity events, between patients with PH who have a low TAPSE and those with a normal TAPSE.

SECONDARY OUTCOMES:
right heart dysfunction | 9 months
  estimate the prevalence of right heart dysfunction in outpatients with pulmonary hypertension in the INCMNSZ
other ultrasound parameters | 9 months
  Show that the presence of pericardial effusion, a right atrial area >34 ml and the presence of septal deviation measured by portable cardiac ultrasound are associated with higher morbidity and mortality events.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutrición Salvador Zubirán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No